CLINICAL TRIAL: NCT04497662
Title: A Phase 1 First-in-human Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Intravenous and Subcutaneous Doses of KPL-404 in Healthy Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of KPL-404 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kiniksa Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kiniksa Pharmaceuticals International, plc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: KPL-404-C101
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KPL-404 (IV Administration) (Experimental)
  Interventions: Drug: KPL-404; Other: Matching Placebo
- KPL-404 (SC Administration) (Experimental)
  Interventions: Drug: KPL-404; Other: Matching Placebo

INTERVENTIONS:
Drug: KPL-404 — humanized IgG4 monoclonal antibody
Other: Matching Placebo — Placebo

SUMMARY:
Phase 1, randomized, double-blind, placebo-controlled first-in-human study to investigate the safety, tolerability, PK and PD properties of single ascending intravenous (IV) and subcutaneous (SC) doses of KPL-404 in healthy subjects

DETAILED DESCRIPTION:
This study includes 2 single ascending dose (SAD) parts; (Part A) IV SAD (up to 5 planned dose level cohorts) and Part B SC SAD (up to 3 planned dose level cohorts).

Safety assessments will include adverse events (AEs), concomitant medications, clinical laboratory, vital signs, 12-lead electrocardiogram, and physical examination. Serial blood samples for PK, PD, and anti-drug antibodies will be performed during each part of the study during the Treatment and Safety Evaluation Period.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy subjects
* Body mass index (BMI) in the range of 18.0 - 32.0 kg/m2

Key Exclusion Criteria:

* Poor peripheral venous access
* Clinically-significant illness within 4 weeks of dose administration
* Active or acute infection requiring systemic antibiotic treatment within 2 weeks prior to Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
TEAEs following IV dosing | Up to 65 days post dose
  After single ascending IV doses, number of subjects with treatment-emergent adverse events (TEAEs) in the KPL-404 dose-level cohorts compared with the (pooled) IV placebo group
TEAEs following SC dosing | Up to 65 days post dose
  After single ascending SC doses, number of subjects with treatment-emergent adverse events (TEAEs) in the KPL-404 dose-level cohorts compared with the (pooled) SC placebo group

CONTACTS AND LOCATIONS:
Locations (2):
- PPD Clinic, Austin, Texas, United States
- Q-Pharm Pty Ltd, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No